CLINICAL TRIAL: NCT01121653
Title: Impact of Oral Magnesium on Neuropathic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0073
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Patient With Neuropathic Pain
Keywords: Neuropathic pain, magnesium
MeSH Terms: conditions — Neuralgia | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Magnogene ® (magnesium) — evaluate on pain scores (neuropathic pain questionnaire and pain numeric scale) and on quality of life, the effect of oral magnesium intake on patients with neuropathic pain comparing with patients receiving placebo,. The study drug will be taken during 4 weeks.

SUMMARY:
Use lay language.

The aim of this study is to evaluate on pain scores (neuropathic pain questionnaire and pain numeric scale) and on quality of life, the effect of oral magnesium intake on patients with neuropathic pain comparing with patients receiving placebo,. The study drug will be taken during 4 weeks.

DETAILED DESCRIPTION:
Protocol description

Visit D0

* patient inclusion after informed signed consent
* clinical exam
* blood sampling (magnesium dosage)
* questionnaires (neuropathic pain and quality of life)
* daily self-evaluation on neuropathic pain scale (Week0 to Week5)

D8 : first intake of study drug (magnesium or placebo)

Visit Week5:

* questionnaires (neuropathic pain and quality of life)
* blood sampling (magnesium dosage)
* clinical exam

ELIGIBILITY:
Inclusion Criteria:

- neuropathic pain

- informed signed consent

Exclusion Criteria:

* magnesium intake contra-indication
* severe renal insufficiency
* quinidine intake
* concomitant treatment change 2weeks before inclusion
* evolutive pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Pain scores (neuropathic pain evaluation questionnaire) | Visit D0

SECONDARY OUTCOMES:
- Numeric scale - quality o f life questionnaires | Visit Week 5

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, MCU-PH, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France